CLINICAL TRIAL: NCT02306161
Title: Randomized Phase 3 Trial Evaluating the Addition of the IGF-1R Monoclonal Antibody Ganitumab (AMG 479, NSC# 750008) to Multiagent Chemotherapy for Patients With Newly Diagnosed Metastatic Ewing Sarcoma
Brief Title: Combination Chemotherapy With or Without Ganitumab in Treating Patients With Newly Diagnosed Metastatic Ewing Sarcoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02380; NCI-2014-02380 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AEWS1221; s15-00442; AEWS1221 (Other: Children's Oncology Group); AEWS1221 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Ewing Sarcoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Neoplasm in the Bone Marrow; Metastatic Malignant Neoplasm in the Lung; Metastatic Peripheral Primitive Neuroectodermal Tumor of Bone; Peripheral Primitive Neuroectodermal Tumor of Soft Tissues
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Cyclophosphamide; Doxorubicin; Etoposide; etoposide phosphate; Congresses as Topic; Radiation; ganitumab; Ifosfamide; Radiosurgery; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A (VDC/IE) (Experimental): See Design Details.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Etoposide Phosphate; Radiation: External Beam Radiation Therapy; Drug: Ifosfamide; Radiation: Stereotactic Radiosurgery; Procedure: Therapeutic Surgical Procedure; Drug: Vincristine; Drug: Vincristine Sulfate
- Regimen B (VDC/IE + ganitumab) (Experimental): INDUCTION THERAPY: Patients receive Induction therapy as in Regimen A and receive ganitumab IV over 30-60 minutes or 60-120 minutes on day 1 of weeks 1, 3, 5, 7, 9, and 11.
  LOCAL CONTROL THERAPY: Between weeks 13-18, patients undergo surgery and/or radiation therapy.
  CONSOLIDATION THERAPY: Patients receive Consolidation therapy as in Regimen A and receive ganitumab IV over 30-60 minutes or 60-120 minutes on day 1 of weeks 7, 9, 11, 13, and 15.
  METASTATIC SITE IRRADIATION: Patients with lung metastases undergo whole lung radiation and patients with bone metastases undergo definitive SBRT or EBRT.
  MAINTENANCE: Patients receive ganitumab IV over 30-60 minutes or 60-120 minutes every 3 weeks for 8 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Etoposide Phosphate; Radiation: External Beam Radiation Therapy; Biological: Ganitumab; Drug: Ifosfamide; Radiation: Stereotactic Radiosurgery; Procedure: Therapeutic Surgical Procedure; Drug: Vincristine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Biological: Ganitumab — Given IV
  Other Names: AMG 479; AMG-479; AMG479; Anti-IGF-1R Human Monoclonal Antibody AMG-479
  Arms: Regimen B (VDC/IE + ganitumab)
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Radiation: Stereotactic Radiosurgery — Undergo SBRT
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Procedure: Therapeutic Surgical Procedure — Undergo surgery
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase III trial studies how well combination chemotherapy with or without ganitumab works in treating patients with newly diagnosed Ewing sarcoma that has spread to other parts of the body. Treatment with drugs that block the IGF-1R pathway, such as ganitumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as vincristine, doxorubicin, cyclophosphamide, ifosfamide, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether adding ganitumab to combination chemotherapy is more effective in treating patients with newly diagnosed metastatic Ewing sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if event-free survival (EFS) in patients with newly diagnosed metastatic Ewing sarcoma treated with multiagent chemotherapy is improved with the addition of ganitumab (AMG 479).

SECONDARY OBJECTIVES:

I. To describe the toxicity of the addition of ganitumab to multimodality therapy for patients with newly diagnosed metastatic Ewing sarcoma.

II. To compare overall survival in patients with newly diagnosed metastatic Ewing sarcoma treated with multiagent chemotherapy with and without the addition of ganitumab.

EXPLORATORY OBJECTIVES:

I. To compare bone marrow response rates in patients with newly diagnosed metastatic Ewing sarcoma treated with multiagent chemotherapy with and without the addition of ganitumab.

II. To describe the toxicity of 6 months of ganitumab monotherapy as maintenance therapy following multimodality therapy in patients with newly diagnosed metastatic Ewing sarcoma.

III. To describe trough levels of ganitumab in a cohort of patients with Ewing sarcoma < 21 years of age treated with 18 mg/kg.

IV. To describe the feasibility of and local failure rates following hypofractionated stereotactic body radiotherapy (SBRT) directed at bone metastases in patients with newly diagnosed metastatic Ewing sarcoma.

V. To determine if EFS, overall survival, bone marrow response rates, and toxicity differ based on serum markers of the insulin-like growth factor 1 (IGF-1) pathway in patients with newly diagnosed metastatic Ewing sarcoma treated with interval compressed chemotherapy with and without the addition of ganitumab.

VI. To determine if EFS, overall survival, and bone marrow response rates differ based on protein, deoxyribose nucleic acid (DNA), and ribonucleic acid (RNA) marker in patients with newly diagnosed metastatic Ewing sarcoma treated with interval compressed chemotherapy with and without the addition of ganitumab.

VII. To evaluate bone marrow micrometastatic disease and tumor cell surface IGF-1R expression at diagnosis and after 3 and 6 cycles of study therapy in patients with newly diagnosed metastatic Ewing sarcoma.

VIII. To determine if the presence of germline polymorphisms in EGFR correlate with response to multiagent therapy with and without ganitumab.

IX. To investigate the ability of fludeoxyglucose F 18-positron emission tomography (FDG-PET) to augment conventional response assessment of primary Ewing sarcoma tumors by magnetic resonance imaging (MRI).

X. To explore FDG-PET response at the primary tumor as a prognostic marker and as a predictive biomarker of clinical activity of IGF-1R inhibition in patients with newly diagnosed metastatic Ewing sarcoma.

XI. To collect data on institutional testing for Ewing sarcoma breakpoint region 1 (EWSR1) translocation status in patients enrolling on study.

XII. To explore the capacity of plasma cell-free DNA analysis to detect tumor-specific genetic changes at initial diagnosis and after initiation of protocol therapy.

XIII. To collect a population of bone marrow metastatic tumor cells by flow cytometry for genomic profiling.

OUTLINE: Patients are randomized to 1 of 2 treatment regimens. (As of 3/20/2019, the study is closed to accrual and patients in Regimen B no longer receive ganitumab.)

REGIMEN A (vincristine sulfate, doxorubicin hydrochloride and cyclophosphamide [VDC] and ifosfamide and etoposide phosphate [IE]):

INDUCTION THERAPY: Patients receive vincristine sulfate intravenously (IV) over 1 minute on day 1, doxorubicin hydrochloride IV over 1-15 minutes on days 1 and 2, and cyclophosphamide IV over 30-60 minutes on day 1 of weeks 1, 5, and 9, and ifosfamide IV over 1 hour on days 1 to 5 and etoposide phosphate IV over 1-2 hours on days 1 to 5 of weeks 3, 7, and 11.

LOCAL CONTROL THERAPY: Between weeks 13-18, patients undergo surgery and/or radiation therapy.

CONSOLIDATION THERAPY: Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1, 7, 9, and 13; doxorubicin hydrochloride IV over 1-15 minutes on days 1 and 2 of weeks 1 and 7, cyclophosphamide IV over 30-60 minutes on day 1 of weeks 1, 7, 9, and 13, ifosfamide IV over 1 hour on days 1 to 5 of weeks 3, 5, 11, and 15, and etoposide phosphate IV over 1-2 hours on days 1 to 5 of weeks 3, 5, 11, and 15.

METASTATIC SITE IRRADIATION: Patients with lung metastases undergo whole lung radiation and patients with bone metastases undergo definitive SBRT or external beam radiation therapy (EBRT).

REGIMEN B (VDC/IE + ganitumab):

INDUCTION THERAPY: Patients receive Induction therapy as in Regimen A and receive ganitumab IV over 30-60 minutes or 60-120 minutes on day 1 of weeks 1, 3, 5, 7, 9, and 11.

LOCAL CONTROL THERAPY: Between weeks 13-18, patients undergo surgery and/or radiation therapy.

CONSOLIDATION THERAPY: Patients receive Consolidation therapy as in Regimen A and receive ganitumab IV over 30-60 minutes or 60-120 minutes on day 1 of weeks 7, 9, 11, 13, and 15.

METASTATIC SITE IRRADIATION: Patients with lung metastases undergo whole lung radiation and patients with bone metastases undergo definitive SBRT or EBRT.

MAINTENANCE: Patients receive ganitumab IV over 30-60 minutes or 60-120 minutes every 3 weeks for 8 cycles.

After completion of study treatment, patients are followed for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic diagnosis (by institutional pathologist) of newly diagnosed Ewing sarcoma or peripheral primitive neuroectodermal tumor (PNET) arising from bone or soft tissue and with metastatic disease involving lung, bone, bone marrow, or other metastatic site
* For the purpose of this study metastatic disease is defined as one or more of the following:

  * Lesions which are discontinuous from the primary tumor, are not regional lymph nodes, and do not share a bone or body cavity with the primary tumor; skip lesions in the same bone as the primary tumor do not constitute metastatic disease; skip lesions in an adjacent bone are considered bone metastases; if there is any doubt whether lesions are metastatic, a biopsy of those lesions should be performed
  * Contralateral pleural effusion and/or contralateral pleural nodules
  * Distant lymph node involvement
  * Patients with pulmonary nodules are considered to have metastatic disease if the patient has:

    * Solitary nodule >= 0.5 cm or multiple nodules of >= 0.3 cm unless lesion is biopsied and negative for tumor
    * Patients with solitary nodule < 0.5 cm or multiple nodules < 0.3 cm are not considered to have lung metastasis unless biopsy documents tumor
  * Bone marrow metastatic disease is based on morphologic evidence of Ewing sarcoma based on hematoxylin and eosin (H&E) stains; in the absence of morphologic evidence of marrow involvement on H&E, patients with bone marrow involvement detected ONLY by flow cytometry, reverse-transcriptase (RT)-polymerase chain reaction (PCR), fluorescence in situ hybridization (FISH), or immunohistochemistry will NOT be considered to have clinical bone marrow involvement for the purposes of this study

    * This study requires bilateral bone marrow biopsies at study entry; the suggested approach for patients with large pelvic tumors in which a posterior iliac crest bone marrow biopsy would track through the tumor is to instead undergo 2 marrow biopsies on the contralateral side (either 2 posterior biopsies or one posterior and one anterior biopsy)
  * Bone metastasis: This study utilizes whole body FDG-PET scans to screen patients for bone metastases; areas suspicious for bone metastasis based on FDG-PET scans require confirmatory anatomic imaging with either MRI or computed tomography (CT) (whole body FDG-PET/CT or FDG-PET/magnetic resonance [MR] scan acceptable); whole body technetium bone scans may be performed at the discretion of the investigator and are not required; for patients without other sites of metastatic disease whose sole metastatic site to qualify for study entry is a single area suspicious for bone metastasis identified by FDG-PET, confirmatory biopsy or anatomic imaging evidence of an associated soft tissue mass at that site is required for study entry
* Patients must have adequate tumor tissue to meet the minimum requirement for submission
* Enrolling institutions are reminded that submission of pre-treatment serum, tumor tissue and whole blood is required
* Patients should only have had a biopsy of the primary tumor without an attempt at complete or partial resection; patients will still be eligible if excision was attempted or accomplished as long as adequate anatomic imaging (MRI for most primary tumor sites) was obtained prior to surgery
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows (performed within 7 days prior to enrollment):

  * Age < 6 months: Maximum serum creatinine (mg/dL): 0.4 for males and females
  * Age 6 months to < 1 year: Maximum serum creatinine (mg/dL): 0.5 for males and females
  * Age 1 to < 2 years: Maximum serum creatinine (mg/dL): 0.6 for males and females
  * Age 2 to < 6 years: Maximum serum creatinine (mg/dL): 0.8 for males and females
  * Age 6 to < 10 years: Maximum serum creatinine (mg/dL): 1 for males and females
  * Age 10 to < 13 years: Maximum serum creatinine (mg/dL): 1.2 for males and females
  * Age 13 to < 16 years: Maximum serum creatinine (mg/dL): 1.5 for males and 1.4 for females
  * Age >= 16 years: Maximum serum creatinine (mg/dL): 1.7 for males and 1.4 for females
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (performed within 7 days prior to enrollment), and
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 3 x upper limit of normal (ULN) for age (performed within 7 days prior to enrollment) (except for patients with liver metastasis who may enroll if ALT < 5 times ULN for age)
* Shortening fraction of >= 27% or
* Ejection fraction of >= 50%
* Patients must have a normal blood sugar level for age to participate; if an initial random draw (ie. non-fasting) blood glucose value is out of range, it is acceptable to repeat this test as a fasting draw
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with regional node involvement as their only site of disease beyond the primary tumor will not be eligible
* Patients whose primary tumors arise in the intra-dural soft tissue (e.g. brain and spinal cord) are not eligible
* Patients who have received prior chemotherapy or radiation therapy are not eligible
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained; lactating females are not eligible unless they have agreed not to breastfeed their infants for the duration of protocol therapy; sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of protocol therapy
* Patients with known pre-existing diabetes mellitus will be excluded from study
* Patients receiving chronic pharmacologic doses of corticosteroids are not eligible; for the purposes of eligibility, chronic exposure is defined as anticipated exposure of > 3 weeks, including the sum of both pre-enrollment and anticipated post-enrollment dosing; patients on acute corticosteroid therapy (=< 3 weeks of total planned exposure) must still meet the normal blood glucose requirement; patients receiving chronic inhaled corticosteroids or chronic physiologic replacement doses of corticosteroids are eligible

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 312 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2026-09-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven G DuBois, Principal Investigator — Children's Oncology Group
Locations (315):
- United States (299):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Onvida Health Yuma Medical Center, Yuma, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] DuBois SG, Krailo MD, Glade-Bender J, Buxton A, Laack N, Randall RL, Chen HX, Seibel NL, Boron M, Terezakis S, Hill-Kayser C, Hayes A, Reid JM, Teot L, Rakheja D, Womer R, Arndt C, Lessnick SL, Crompton BD, Kolb EA, Daldrup-Link H, Eutsler E, Reed DR, Janeway KA, Gorlick RG. Randomized Phase III Trial of Ganitumab With Interval-Compressed Chemotherapy for Patients With Newly Diagnosed Metastatic Ewing Sarcoma: A Report From the Children's Oncology Group. J Clin Oncol. 2023 Apr 10;41(11):2098-2107. doi: 10.1200/JCO.22.01815. Epub 2023 Jan 20. PMID 36669140
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A (VDC/IE): INDUCTION THERAPY: Patients receive Induction therapy with alternating cycles of VDC and IE given every 2 weeks for 6 cycles.
  LOCAL CONTROL THERAPY: Between weeks 13-18, patients undergo surgery and/or radiation therapy.
  CONSOLIDATION THERAPY: Patients receive Consolidation therapy with alternating cycles of VDC and IE given every 2 weeks for 8 cycles.
  METASTATIC SITE IRRADIATION: Patients with lung metastases undergo whole lung radiation and patients with bone metastases undergo definitive SBRT or EBRT.
  Cyclophosphamide: Given IV
  Doxorubicin: Given IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Etoposide Phosphate: Given IV
  External Beam Radiation Therapy: Undergo EBRT
  Ifosfamide: Given IV
  Stereotactic Radiosurgery: Undergo SBRT
  Therapeutic Surgical Procedure: Undergo surgery
  Vincristine: Given IV
  Vincristine Sulfate: Given IV
- Regimen B (VDC/IE + Ganitumab): INDUCTION THERAPY: Patients receive Induction therapy as in Regimen A and receive ganitumab IV over 30-60 minutes or 60-120 minutes on day 1 of weeks 1, 3, 5, 7, 9, and 11.
  LOCAL CONTROL THERAPY: Between weeks 13-18, patients undergo surgery and/or radiation therapy.
  CONSOLIDATION THERAPY: Patients receive Consolidation therapy as in Regimen A and receive ganitumab IV over 30-60 minutes or 60-120 minutes on day 1 of weeks 7, 9, 11, 13, and 15.
  METASTATIC SITE IRRADIATION: Patients with lung metastases undergo whole lung radiation and patients with bone metastases undergo definitive SBRT or EBRT.
  MAINTENANCE: Patients receive ganitumab IV over 30-60 minutes or 60-120 minutes every 3 weeks for 8 cycles.
  Cyclophosphamide: Given IV
  Doxorubicin: Given IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Etoposide Phosphate: Given IV
  External Beam Radiation Therapy: Undergo EBRT
  Ganitumab: Given IV
  Ifosfamide: Given IV
  Stereotactic Radiosurgery: Undergo SBRT
  Therapeutic Surgical Procedure: Undergo surgery
  Vincristine: Given IV
  Vincristine Sulfate: Given IV
Period: Overall Study
Arm/Group | Regimen A (VDC/IE) | Regimen B (VDC/IE + Ganitumab)
Started | 157 | 155
Completed | 93 | 86
Not Completed | 64 | 69
Not completed — Death | 1 | 3
Not completed — Lack of Efficacy | 20 | 43
Not completed — Physician Decision | 30 | 18
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Ineligible | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (VDC/IE) | Regimen B (VDC/IE + Ganitumab) | Total
Number analyzed (Participants) | 157 | 155 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 124 | 123 | 247
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 14.89 [11.47 to 18.09] | 15.16 [11.32 to 18.11] | 15.03 [11.32 to 18.09]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 69 | 140
  Male | 86 | 86 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 23 | 51
  Not Hispanic or Latino | 113 | 116 | 229
  Unknown or Not Reported | 16 | 16 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 5 | 3 | 8
  White | 128 | 125 | 253
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 17 | 21 | 38
Region of Enrollment [Number; unit: participants]
  United States | 144 | 142 | 286
  Canada | 10 | 11 | 21
  China | 0 | 1 | 1
  Guatemala | 1 | 0 | 1
  Puerto Rico | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Estimated 5-year EFS where EFS is calculated as the time from study enrollment to disease progression, disease relapse, occurrence of a second malignant neoplasm, death from any cause or last follow-up whichever occurs first. Kaplan-Meier method is used for estimation. Patients without an event are censored at last contact.
Time Frame: 5 years after enrollment
Population: Only eligible patients are considered in the calculation of this outcome measure.
Measure: Number (95% Confidence Interval); unit: percent probability of participants
Arm/Group | Regimen A (VDC/IE) | Regimen B (VDC/IE + Ganitumab)
Number analyzed (Participants) | 148 | 150
percent probability of participants | 30.88 [22.50 to 39.63] | 30.4 [22.40 to 38.88]

2. Secondary Outcome: Overall Survival
Description: Time from study enrollment to death or last patient contact.
Time Frame: 5 years after enrollment
Population: Only eligible patients are considered in the calculation of this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Regimen A (VDC/IE) | Regimen B (VDC/IE + Ganitumab)
Number analyzed (Participants) | 148 | 150
Percent Probability | 44.93 [33.61 to 55.60] | 48.19 [38.15 to 57.52]

3. Secondary Outcome: Frequency of Toxicity-events
Description: The number of induction or consolidation reporting periods in which a CTC version 4 codeable grade 4 or greater non-hematological adverse event, grade 3 or greater left ventricular systolic dysfunction or the reporting period is terminated because of a CTC codeable event.
Time Frame: Up to 202 days
Population: Only eligible patients who received at least one dose of assigned protocol therapy are considered in the calculation of this outcome measure. Five hundred twenty-seven (527) reporting periods were contributed by patients enrolled on Regimen A; Five hundred seventy-six 576 reporting periods were contributed by patients enrolled on Regimen B.
Measure: Number; unit: Reporting Periods
Units Other Than Participants: Reporting Periods
Arm/Group | Regimen A (VDC/IE) | Regimen B (VDC/IE + Ganitumab)
Number analyzed (Participants) | 145 | 150
Number analyzed (Reporting Periods) | 527 | 576
Reporting Periods | 10 | 27

4. Other Pre Specified Outcome: Serum IGF Pathway Component and Tissue Protein, Deoxyribonucleic Acid (DNA), and Ribonucleic Acid Markers
Description: In addition to the log rank test the modeling approach will be used for the primary study comparison. Linear trend in EFS-risk will be investigated by segregating the marker level according to quartiles. For bone marrow response rate analyses, Fisher's exact test will be used to compare the objective bone marrow response rate (complete response vs. incomplete response) at start of local control between patients with biomarker levels above and below the group median.
Time Frame: Up to 10 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Tumor Cell Surface IGF-1R Expression
Description: Extent of tumor cell IGF-1R co-expression will also be reported. Change in tumor cell IGF-1R co-expression in patients treated with and without ganitumab will be reported descriptively.
Time Frame: Up to 307 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Germline Polymorphisms in EGFR
Description: EFS will be compared between patients with and without the presence of the minor allele using the log rank test, both for the entire patient population and for patients randomized to ganitumab.
Time Frame: Up to 10 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: EWS Translocation
Description: The institutional result of EWS tumor testing will be categorized as translocation detected (yes v. no) and the type of translocation detected will also be recorded. The proportion of patients with a particular EWS translocation variant will be tabulated.
Time Frame: Up to 10 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Circulating Tumor DNA (ctDNA) Testing
Description: Will report the proportion of patients that have a change in translocation result associated with ctDNA testing across time periods.
Time Frame: Up to 202 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Serial Genomic Profiling
Description: Will be identified by flow cytometry. Profiles will be presented graphically, and samples obtained from different sites of tumor within the same individual will also be presented.
Time Frame: Up to 307 days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Occurrence of Sinusoidal Obstructive Disease (SOS) Associated With the Addition of Ganitumab to VDC/IE
Description: The number of induction and maintenance cycles received by patients randomized to the experimental therapy where SOS is observed. Only patients who receive all reporting period therapy or experience SOS will contribute to this outcome measure.
Time Frame: Up to 202 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Frequency of Resolution of Bone Marrow Metastases
Description: The number of patients who are enrolled with bone marrow metastases whose bone marrow disease is not detected after evaluation at the time of of first local control measure or the end of the Induction reporting period, whichever comes first. Only eligible patients who receive at least one dose of randomized treatment assignment will be considered for this measure.
Time Frame: Up to 84 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Frequency of Toxicity Events During Ganitumab Maintenance
Description: The number of induction or consolidation reporting periods in which a CTC version 4 codeable non-hematological adverse event, grade 3 left ventricular systolic dysfunction or the reporting period is terminated because of a CTC codeable event.
Time Frame: Up to 307 days
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Trough Levels of Serum Ganitumab
Description: Trough levels of serum ganitumab prior to the second dose of ganitumab during induction obtained will be categorized as less than 10 micrograms per milliliter or greater than or equal to 10 micrograms per milliliter. This analysis will be conducted for the first 10 eligible patients who receive ganitumab.
Time Frame: Up to 15 days
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Proportion of Patients Who Successfully Receive Planned Stereotactic Body Radiotherapy (SBRT)
Description: A patient who has SBRT planned for at least one metastatic site and receives successful SBRT treatment to at least 85% of metastatic sites in the treatment plan. Successful treatment is determined by IROC review criteria. Only eligible patients start the metastatic site radiation reporting period will be considered for this outcome measure.
Time Frame: 202 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored up to 358 days from study enrollment, All-Cause Mortality monitored up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients and those who did not receive therapy are excluded. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Regimen A (VDC/IE) | Regimen B (VDC/IE + Ganitumab)
All-Cause Mortality (participants affected / at risk) | 61/145 | 67/150
Serious Adverse Events (participants affected / at risk) | 3/145 | 45/150
Other Adverse Events (participants affected / at risk) | 114/145 | 122/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (VDC/IE) (N=145) | Regimen B (VDC/IE + Ganitumab) (N=150)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 9 (9)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6)
Fever (General disorders) | 1 (1) | 2 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 0 (0) | 2 (2)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (VDC/IE) (N=145) | Regimen B (VDC/IE + Ganitumab) (N=150)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 7 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 38 (38) | 50 (50)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (6) | 9 (9)
Nausea (Gastrointestinal disorders) | 8 (8) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4) | 6 (6)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 2 (2)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 26 (26) | 20 (20)
Neutrophil count decreased (Investigations) | 91 (91) | 92 (92)
Platelet count decreased (Investigations) | 24 (24) | 68 (68)
Weight loss (Investigations) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 82 (82) | 85 (85)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT02306161/Prot_SAP_000.pdf